CLINICAL TRIAL: NCT02706184
Title: Randomized, Placebo Controlled Phase III Trial of a Microbiological Concomitant Therapy/Prevention of Chemotherapeutical Induced Diarrhea (Caused by Inflammation and an Impaired Intestinal Barrier) With E. Coli Nissle 1917 (EcN)-Suspension in Patients With Gastric and Colorectal Cancer
Brief Title: E. Coli Nissle in Oncology
Acronym: EcNO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: Ardeypharm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZKES-EcNO-2015
Record Dates: First submitted 2016-02-23; First posted 2016-03-11 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Gastric Cancer; Colorectal Cancer
Keywords: gastric cancer; colorectal cancer; chemotherapy induced diarrhea; 5-Fluoruracil; chemotherapeutic remedy
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients receive E. coli Nissle suspension
  Interventions: Drug: E. coli Nissle suspension
- Control (Placebo Comparator): Patients receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E. coli Nissle suspension — Patients receive E. coli Nissle suspension
  Other Names: Mutaflor Suspension®
  Arms: Intervention
Drug: Placebo — Placebo
  Arms: Control

SUMMARY:
In patients with gastric or colorectal cancers, where a treatment with 5-Fluoruracil in combination with other chemotherapeutic remedies (FLO, FOLFOX, FOLFOX-Bev, FOLFIRI) is planned, it shall be investigated whether E. coli Nissle suspension has an effect on duration and intensity of chemotherapy induced diarrhea.

DETAILED DESCRIPTION:
Chemotherapy is used frequently for treating tumors. For many kinds of tumors, chemotherapy is an effective way of treatment. Besides the desired effects on neoplastic cells, the cytotoxic effects often lead to undesirable effects in other cells. Particularly the epithelial tissue of the gastrointestinal tract is affected, mucositis and diarrhea occur. By loss of water and electrolytes, diarrhea often make delay in chemotherapy necessary. Besides mucositis, a chemotherapy also causes changes in gut microbiota as animal models proof. It is well known, than probiotics shorten diarrhea. So far, the use of probiotics in chemotherapy patients was only investigated in one single study. Severity of diarrhea was reduced compared to placebo. Escherichia coli Nissle 1917 (EcN) is a well investigated probiotic. In cell culture, the supernatant of EcN reduced the noxious effect of 5-Fluoruracil concerning cell toxicity and disruption of barrier function.

Therefore, the aim of this study is whether in patients with gastric or colorectal cancers, where a treatment with 5-Fluoruracil in combination with other chemotherapeutic remedies (FLO, FOLFOX, FOLFOX-Bev, FOLFIRI) is planned, EcN-Suspension is capable to reduce duration and intensity of chemotherapy induced diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults
* patients with gastric or colorectal cancer (stages III or IV), where a treatment with 5-Fluoruracil in combination with other chemotherapeutic remedies (FLO, FOLFOX, FOLFOX-Bev, FOLFIRI) is planned
* life expectancy of at least the trial duration
* the first administering of the product under investigation must be able to take place 72 hours before or after the beginning of the chemotherapeutical treatment, ideally at the same time
* an inclusion into the study is only possible at the beginning of the first chemotherapeutic cycle
* fertile female patients (aged 49 years or minor, the last menstruation occured in less than two years) have to be either surgically sterilized or use the same highly effective method of contraception for at least three months
* willingness to refrain from other probiotics or probiotic yoghurts, a systematic change of eating behavior should not be planned
* sufficient knowledge of german language and sufficient psychological state for being able to answer questionnaires and assessment scales
* informed written consent

Exclusion Criteria:

* Participation in other clinical trials (currently or within the last 30 days)
* intolerance against ingredients of the product under investigation
* pregnancy or lactation
* being not able to consume the product under investigation orally
* antidiarrheal therapy with antibiotics
* alcohol or drug abuse within the last six months
* any health condition (including abnormal blood parameters) which refuses a patient from taking part in the study according to the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Common toxicity criteria for diarrhea Version 4.0 | Baseline vs. week 12

SECONDARY OUTCOMES:
Quality of life by SF-12 questionnaire | Baseline vs. week 12
Quality of life by FACIT-D questionnaire | Baseline vs. week 12
stool consistency by Bristol stool scale | Baseline vs. week 12
Body mass index in kg/m^2 | Baseline vs. week 12
Phase angle | Baseline vs. week 12
C-reactive protein | Baseline vs. week 12
Hematocrit | Baseline vs. week 12
alpha-1-Antitrypsin | Baseline vs. week 12
Calprotectin | Baseline vs. week 12
Body cell mass in kg | Baseline vs. week 12
ECM/BCM-Index | Baseline vs. week 12
  ECM = extracellular mass BCM = body cell mass

OTHER OUTCOMES:
stool water content | Baseline vs. week 12
stool microbiome analyses | Baseline vs. week 12

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C. Bischoff, Prof., Study Director — ZKES GmbH
Locations (4):
- Germany (4):
  - Klinikum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg
  - Paracelsus-Krankenhaus Ruit, Ostfildern, Baden-Wurttemberg
  - Klinikum am Steinenberg /Ermstalklinik, Reutlingen, Baden-Wurttemberg
  - Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg

IPD SHARING:
Plan to Share IPD: No